CLINICAL TRIAL: NCT05292768
Title: Are Mast Cells Involved in Autoinflammatory Diseases
Acronym: INFLAMAST
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Imagine (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP210126
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Autoinflammatory Disease; FMF; TRAPS; MKD; Cryopyrin Associated Periodic Syndrome; Haploinsufficiency
Keywords: Autoinflammatory disease; Mast cells; Mast cell activation syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Mast Cell Activation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples Digestive, renal or cutaneous biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with AID
- Control patients with mastocytosis
- Control patients with normal digestive biopsy
- Control patients with renal biopsy
- Control patients with inflammatory disease
- Healthy control from healthcare workers

SUMMARY:
Autoinflammatory diseases (AID) are caused by innate immunity dysregulation. AID pathophysiology is only partly understood, especially in the case of unclassified AID. Mast cells (MC) are innate immune cells associated with a spectrum of disease between systemic mastocytosis and mast cell activation syndrome. The implication of MC has been shown in cryopyrin associated periodic syndrome (CAPS).Our aim is to evaluate the involvement of MC in AID by assessing clinical and biological signs of MC activation and studying cutaneous and digestive biopsies.

DETAILED DESCRIPTION:
Autoinflammatory diseases (AID) are caused by innate immunity dysregulation and characterized by recurrent bouts of fever, frequently associated with digestive, articular or cutaneous symptoms, and sometimes ocular, auricular or neurologic inflammation. The most frequent monogenic AID is Familial Mediterranean fever (FMF).

Despite recent genetic progress AID pathophysiology is only partly understood, especially in the case of unclassified AID.

Mast cells (MC) are innate immune cells associated with a spectrum of disease between systemic mastocytosis and mast cell activation syndrome (MCAS). In MCAS, patients have various symptoms including abdominal pain, bloating, pruritus, flush, anxiety, fatigue, among which some are similar to those seen in patients with AID. The implication of MC has been shown in cryopyrin associated periodic syndrome (CAPS).

Our hypothesis is that MC could be involved in AID pathophysiology,

In order to test this hypothesis, we plan to study :

* clinical MC activation symptoms via a standardized clinical score
* biological MC mediators : by measuring total serum tryptase and histamine in total blood, plasma and urine
* MC infiltration on gastro-intestinal (GI) tract and cutaneous biopsies We will compare clinical MC activation score in AID patients to patients with mastocytosis, with other inflammatory diseases, and with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with Auto-inflammatory diseases already followed up at the CeRéMAIA (french national reference center for autoinflamamtory diseases and AA amyloidosis) of Tenon hospital and included in the JIRcohorte
* Healthy adult controls, age- and sex-matched with MAI patients, and controls with mastocytosis, an immuno-inflammatory disease.
* Subject affiliated to or entitled to a social security scheme
* Collection of the patient's or healthy control's non-opposition

Exclusion Criteria:

* Subjects unable to answer questions or express themselves
* Subjects who do not speak French
* Subject deprived of liberty or under legal protection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients wil be recruited in tertiary university centres of the Assitance Publique des Hopitaux de Paris.
  Healthy controls will be recruited from volunteer healthcare workers in Assitance Publique des Hopitaux de Paris
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
: presence of MCAS | at inclusion
  presence of clinical and biological markers of MCAS

SECONDARY OUTCOMES:
comparison of clinical symptoms of MC activation between groups | at inclusion
  we will compare clinical symptoms of MC activation between AID patients and other groups
MC mediators associated to AID | at inclusion
  determine which MC mediators are elevated in AID and if they correlate with inflammation
MC infiltration in biopsies from AID patients | at inclusion, retrospectively
  we will study MC infiltration in digestive, renale and cutaneous biopsies from patients with AID and compare them with biopsies from the other groups from subgroups of patients who had a biopsy performed.
basophilic polynuclear activation in AID patients | at inclusion, retrospectively
  we will study basophilic polynuclear activation from blood samples of AID patients

CONTACTS AND LOCATIONS:
Overall Officials: Sophie GEORGIN-LAVIALLE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Interne, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided